CLINICAL TRIAL: NCT07101705
Title: An Open-label, Single-arm Clinical Study to Evaluate the Safety and Preliminary Efficacy of OriV508 Injection in Treating Relapsed/Refractory Hematological Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: OriCell Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, MEI HENG, Professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OriV508-T1
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma (MM); Non-Hodgkin Lymphoma (NHL)
Keywords: BCMA/CD19; multiple myeloma; Non-Hodgkin lymphoma; In vivo CAR-T
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OriV508 injection (Experimental): OriV508 injection is one kind of non-replicative self-inactivating lentivirus vector which carries an effective BCMA/CD19 dual-target CAR. OriV508 can be administered intravenously and produce BCMA/CD19 CAR-T in vivo.
  Interventions: Drug: OriV508 Injection

INTERVENTIONS:
Drug: OriV508 Injection — OriV508 injection is one kind of non-replicative self-inactivating lentivirus vector which carries an effective BCMA/CD19 dual-target CAR. OriV508 can be administered intravenously and produce BCMA/CD19 CAR-T in vivo.
  Other Names: OriV508

SUMMARY:
This is a single center, single arm, open-label, dose escalation, phase 1 study to evaluate the safety, tolerability, preliminary efficacy and immunogenicity of OriV508 injection for patients with relapsed/refractory hematological malignancies.

DETAILED DESCRIPTION:
This investigator-initiated clinical study aims to evaluate OriV506 injection, the self-inactivating lentiviral vector that carries a BCMA/CD19 dual-target CAR, in patients with relapsed refractory B-cell hematological malignancies. The study employs a dose-escalation design to assess safety, tolerability, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 75 years.
2. ECOG scores 0-1.
3. Expected survival time ≥ 12 weeks.
4. Have a record of confirmed multiple myeloma (MM) according to IMWG criteria, or a record of histologically confirmed aggressive B-cell non-Hodgkin lymphoma (B-NHL). According to the definition of the 2022 World Health Organization (WHO) classification, the pathological types of aggressive B-NHL include: diffuse large B-cell lymphoma, not otherwise specified; diffuse large B-cell lymphoma/high-grade B-cell lymphoma with MYC and BCL2 rearrangements; high-grade B-cell lymphoma, not otherwise specified; primary mediastinal B-cell lymphoma; mantle cell lymphoma; grade 3b follicular lymphoma; large B-cell lymphoma transformed from indolent B-NHL.
5. For MM subjects only: (1) Have received at least 2 lines of anti-tumor therapy, with each line of therapy undergoing at least one complete treatment cycle, and have experienced disease progression during or within 12 months after the last treatment; or be judged by the investigator as double-refractory to immunomodulators and proteasome inhibitors, and did not achieve a minimal response (MR) or better during the last treatment or experienced disease progression within 60 days after the end of treatment. (2) Have measurable lesions during the screening period, meeting any of the following criteria: (a) Serum M-protein ≥ 0.5 g/dL; (b) Urine M-protein≥ 200 mg/24h; (c) Involved free light chain (FLC) level ≥10 mg/dL provided serum FLC ratio is abnormal; (d) Plasma cell percentage ≥30% detected by bone marrow aspirate/biopsy; (e) Presence of at least one extramedullary lesion with a maximum diameter ≥ 2 cm.
6. For aggressive B-NHL subjects only: (1) Have received at least 2 lines of anti-tumor therapy, and are refractory to the last line of therapy (at least 2 cycles) (best response is PD or SD) or have experienced disease progression after the end of treatment. Previous treatments must include standard treatment regimens with anti-CD20 monoclonal antibodies (except for subjects with CD20-negative tumors) and anthracyclines; (2) Have at least one measurable lesion during the screening period: lymph node lesions must have a longest diameter > 1.5 cm, and extranodal lesions must have a longest diameter > 1.0 cm.
7. Hemogram meets the following requirements:

   * Hemoglobin ≥ 6 g/dL (no red blood cell transfusion within 1 week prior to screening, recombinant human erythropoietin is permitted);
   * Absolute neutrophil count (ANC) ≥ 750 /μL (no granulocyte colony-stimulating factor (G-CSF) used within 1 week prior to screening or no pegylated G-CSF used within 2 weeks prior to screening);
   * Platelet count ≥ 50,000 /μL;
   * Lymphocyte count ≥ 500 /μL.
8. Renal function: Creatinine clearance (CrCl) (Modification of Diet in Renal Disease (MDRD) formula) ≥ 40 mL/min/1.73m² (for MM subjects with CrCl < 40 mL/min/1.73m², the investigator can decide whether to enroll based on clinical indications).
9. Liver function: Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3.0 × upper limit of normal (ULN), total bilirubin ≤ 1.5 × ULN (for subjects with Gilbert's syndrome or liver invasion by tumor, ALT and AST ≤ 5.0 × ULN and total bilirubin ≤ 3 × ULN are permitted).
10. Cardiac function: Left ventricular ejection fraction ≥ 45%.
11. Pulmonary function: Pulse oxygen saturation ≥ 92% without oxygen inhalation.
12. Women with childbearing potential must have a negative blood pregnancy test and not be in the lactation period.
13. Men and women with childbearing potential must agree to use effective contraceptive measures from the time of signing the informed consent form (ICF) until 1 year after the investigational drug administration.
14. Men and women with childbearing potential must agree not to donate reproductive cells such as sperm or eggs (oocytes) from the time of signing the ICF until 1 year after the investigational drug administration.
15. The participant or their legally authorized representative agrees to participate in this clinical trial and signs the ICF, indicating that he/she understands the objective and procedures of this clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. The subject has received the following therapy prior to signing the ICF:

   * Small molecule targeted therapy, epigenetic therapy, or treatment with an investigational drug or used an invasive investigational medical device within 14 days or at least 5 half-lives, whichever is longer;
   * Immunosuppressive agent therapy (such as tacrolimus, mycophenolate mofetil, etc.) within 28 days;
   * Monoclonal antibody treatment within 21 days;
   * Cytotoxic therapy within 14 days;
   * Proteasome inhibitor therapy within 14 days;
   * Immunomodulator agent therapy within 7 days;
   * Therapeutic dose of corticosteroids (defined as prednisone ≥ 20 mg/day or equivalent dose of other corticosteroids) within 72 hours, but physiological replacement dose, topical and inhaled corticosteroids are permitted;
   * Radiotherapy within 28 days (only for subjects whose radiation field covers > 5% of bone marrow reserve).
2. Received autologous hematopoietic stem cell transplantation within 24 weeks prior to signing the ICF.
3. Received organ transplantation or allogeneic hematopoietic stem cell transplantation.
4. Have other malignant tumors prior to screening, except for the following cases: malignant tumors that have received radical treatment and have no known active disease within 2 years prior to screening; or adequately treated non-melanoma skin cancer with no evidence of active disease.
5. Previously treated with any viral therapy using vesicular stomatitis virus G (VSVG)-pseudotyped virus.
6. Known active central nervous system involvement or clinical signs of meningeal involvement.
7. Complicated with severe uncontrolled active infections (bacterial, viral, fungal, etc.).
8. Have active autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) or diseases requiring systemic application of immunosuppressive drugs.
9. Have hereditary bleeding/coagulation diseases, other diseases that may increase the risk of bleeding, etc.
10. Have active deep vein thrombosis (cancer emboli or thrombus) or pulmonary embolism within 12 weeks prior to signing the ICF, but if the investigator judges that the thrombus has been clinically treated and has no risk of detachment, enrollment is permitted.
11. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA titer exceeding the normal range; positive for hepatitis C virus (HCV) antibody with peripheral blood hepatitis C virus (HCV) RNA titer exceeding the normal range; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis test.
12. Complicated with symptomatic heart failure or other severe cardiac diseases such as arrhythmia:

    * New York Heart Association (NYHA) class III or IV congestive heart failure;
    * Myocardial infarction, coronary artery bypass grafting (CABG) or coronary stent implantation within 24 weeks prior to signing the ICF;
    * Clinically significant ventricular arrhythmia, or history of unexplained syncope (except those caused by vasovagal or dehydration);
    * Significant non-ischemic cardiomyopathy history.
13. Have other clinically significant diseases, including:

    * Primary immunodeficiency;
    * Stroke or epileptic seizure within 24 weeks prior to signing the ICF;
    * Obvious clinical evidence of dementia or mental status changes;
    * History of Parkinson's disease or Parkinson-like movement disorders.
14. Underwent surgery within 2 weeks prior to signing the ICF or plan to undergo surgery within 2 weeks after drug administration, except for surgery under local anesthesia.
15. Used attenuated/inactivated vaccines within 28 days prior to signing the ICF.
16. Known severe allergic reaction to OriV508 or its formulation components.
17. Known severe allergic reaction to tocilizumab.
18. Inability to establish venous access.
19. Other situations deemed unsuitable for participating in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Dose-limiting toxicities (DLTs) are evaluated between the infusion and 28 days post-infusion.
Cytokine release syndrome (CRS) | up to Day 28 post-infusion
  Cytokine release syndrome (CRS) would be graded according to the ASTCT consensus.
Immune cell-associated immune effector cell-associated neurotoxicity syndrome (ICANS) | up to Day 28 post-infusion
  ICANS would be scored according to Immune Effector Cell-Associated Encephalopathy (ICE), and then graded by the ASTCT consensus.
Treatment-associated adverse effects (AEs) | From the enrollment to up to the end of treatment at 96 weeks after treatment of OriV508 or withdrawal from the study
  All other AEs would be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate (ORR) | From OriV508 infusion to the end of treatment at 96 weeks
  Clinical efficacy of MM cohort can be evaluated according to the 2016 International Myeloma Working Group consensus criteria. ORR = stringent complete response (sCR) rate + complete response (CR) rate + very good partial response (VGPR) rate + partial response (PR) rate.
  Clinical efficacy of B-NHL cohort can be evaluated according to the Lugano 2014 criteria. ORR = CR+PR.
Complete response (CR) rate | From OriV508 infusion to the end of treatment at 96 weeks
  Clinical efficacy of MM cohort can be evaluated according to the 2016 International Myeloma Working Group consensus criteria.Clinical efficacy of B-NHL cohort can be evaluated according to the Lugano 2014 criteria.
Duration of response (DOR) | From OriV508 infusion to the end of the treatment at 96 weeks
  DOR is defined as the interval between the first sCR, CR, VGPR, or PR after infusion and the disease progression or death.
Time to response (TTR) | From OriV508 infusion to the end of treatment at 96 weeks
  TTR is defined as the interval between the initiation of OriV508 treatment and the first assessment of sCR, CR, VGPR or PR.
Progression-free survival (PFS) | From OriV508 infusion to the end of the treatment at 96 weeks
  PFS is defined as the interval between a subject's receipt of OriV508 infusion and the first assessment of disease progression or death.
Overall survival (OS) | From OriV508 infusion to the end of treatment at 96 weeks
  OS is defined as the interval between a subject's receipt of OriV508 infusion and death from any cause.
Minimal residual disease (MRD) - negative assessment | From OriV508 infusion to the end of treatment at 96 weeks
  This outcome is primarily chosen for patients with multiple myeloma and aims to calculate the proportion of all patients achieving MRD negative status.
CAR-T kinetics | Baseline, Day 4, Day 7, Day 10, Day 14, Day 21, Day 28, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 or withdrawal from the study
  CAR-T kinetics would be detected by flow cytometry and droplet digital or quantitative polymerase chain reaction in peripheral blood and bone marrow at each important time points. Cmax is the peak expansion value of CAR-T cells.

OTHER OUTCOMES:
Immunogenicity of OriV508 injection | up to 96 weeks post-infusion
  Anti-drug antibody (ADA) would be detected by ELISA or FCM.
Replication competent lentivirus (RCL) | Baseline, Week 12, Week 24, Week 48, Week 96 post-infusion or withdrawal from the study.
  RCL refers to a lentivirus (usually genetically unmodified) that retains the ability to autonomously replicate and produce infectious viral particles in host cells.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Ph.D&M.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No